CLINICAL TRIAL: NCT07393464
Title: The Efficacy and Safety of Pyrroloquinoline Quinone add-on Treatment for Negative and Cognitive Symptoms in Chronic Schizophrenia
Brief Title: PQQ for Cognitive and Negative Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Principal Investigator, Yang Chenghao, PhD, Tianjin Anding Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJPQQ2026
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Cognitive Symptoms; Negative Symptoms
Keywords: cognitive symptom; negative symptom; schizophrenia; Pyrroloquinoline Quinone; MCCB
MeSH Terms: conditions — Schizophrenia; Neurobehavioral Manifestations | interventions — PQQ Cofactor; Dietary Fiber

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to receive either PQQ or a matched placebo in a double-blind, randomized controlled design. Treatment allocation will remain concealed from investigators, clinicians, and statisticians until the completion of data analysis. To ensure blinding, the placebo is matched to PQQ in appearance, odor, and color, and both are dispensed in identically sealed bottles. Each bottle is labeled as trial medication and assigned a random code (1-70) by the trial pharmacist, who maintains exclusive access to the randomization list stored securely until study completion. An independent individual, not involved in any aspect of the trial, generates the random allocation sequence based on the sequential enrollment of participants. Participants are assigned to either the intervention or control group according to this randomization protocol, using a table of random numbers. Participants are interviewed individually to prevent communication about treatment experiences. Medicat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PQQ group (Experimental)
  Interventions: Dietary Supplement: Pyrroloquinoline quinone (PQQ)
- Control group (Placebo Comparator)
  Interventions: Dietary Supplement: placebo (dietary fiber)

INTERVENTIONS:
Dietary Supplement: Pyrroloquinoline quinone (PQQ) — Patients with chronic schizophrenia in experimental group will take 20 mg of PQQ orally every day for a total of 12 weeks.
  Arms: PQQ group
Dietary Supplement: placebo (dietary fiber) — Patients with chronic schizophrenia in control group will a capsule of placebo orally every day for a total of 12 weeks.
  Arms: Control group

SUMMARY:
Schizophrenia is a complex mental disorder characterized by a range of symptoms, including negative symptoms and cognitive impairments. Recent research has indicated the potential benefits of targeting mitochondrial dysfunction, oxidative stress, and inflammatory responses in alleviating symptoms of schizophrenia. However, the results remain inconsistent across various studies. This study aims to evaluate the efficacy of Pyrroloquinoline quinone (PQQ) in reducing negative symptoms and improving cognitive function in patients with chronic schizophrenia. The investigation will focus on changes in severity scores from baseline to endpoint, as well as during an eight-week follow-up period. A double-blind, randomized controlled trial will be conducted involving participants diagnosed with chronic schizophrenia. Participants will be randomly assigned to receive either PQQ or a matched placebo. Data will be collected through questionnaires and neuroimaging techniques, including resting-state scans and multimodal tasks to assess functional connectivity and activation in target brain regions. Statistical analyses will include descriptive statistics, voxel-by-voxel multiple regression, and linear mixed models to account for repeated measurements. Additionally, potential moderating effects of demographic factors such as age and gender will be examined using ANCOVAs. The study will also monitor adverse events and ensure participant safety through a rigorous reporting and unblinding procedure. It is hope to provide insights into the therapeutic potential of PQQ in managing schizophrenia symptoms, contributing to the development of more effective treatment strategies for this challenging condition.

ELIGIBILITY:
Inclusion criteria:

Eligible male and female patients aged 18 to 50 years, diagnosed with schizophrenia according to the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5), will be included in the study. Participants are required to meet the following criteria: a Positive and Negative Syndrome Scale (PANSS) total scores of ≥ 60 (indicating an active phase of the illness), a PANSS negative subscale scores of ≥ 20, and a duration of illness of at least 2 years (indicating chronic schizophrenia). Additionally, participants must have been on a stable dose of antipsychotic medication for a minimum of 6 weeks prior to enrollment, and the use of antioxidants or anti-inflammatory medications is prohibited within 2 weeks preceding enrollment.

Exclusion criteria:

Patients with comorbid psychiatric disorders as defined by the DSM-5, such as substance abuse or dependence (excluding nicotine), or intellectual disability (IQ < 70); those with significant depressive symptoms, defined as a score ≥14 on the 17-item Hamilton Depression Rating Scale (HAMD-17) or ≥ 4 on the depression item of PANSS; individuals with severe medical or neurological conditions, or those unable to communicate effectively; patients with a known allergy to PQQ disodium salt, or who are pregnant, breastfeeding, or have severe hepatic or renal impairment; women of childbearing potential who are not using reliable contraception; patients who have received modified electroconvulsive therapy (MECT) or other physical treatments within six months prior to enrollment; and those currently receiving treatments that cannot be discontinued, including antidepressants, mood stabilizers, antihistamines, or combination therapy with two or more antipsychotics (except for low-dose aripiprazole, ≤ 5 mg/day, used solely for prolactin reduction).

Additional exclusion criteria for participants undergoing fMRI scanning:

Participants are required to complete a comprehensive safety questionnaire addressing potential risks associated with exposure to a 3-Tesla magnetic field and the MRI environment. MRI-specific exclusion criteria include: the presence of MRI-incompatible implants (e.g., cochlear implants, insulin pumps, pacemakers, or other metallic implants); a history of possible intraocular metallic foreign bodies due to manual labor without appropriate eye protection; tattoos containing red pigments; claustrophobia; or unwillingness to be informed of any incidental structural brain abnormalities detected during the scan.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
cognitive symptoms | From enrollment to the end of 12 weeks
  the changes in scores of MCCB between the baseline and the first post-treatment measurement.
negative symptoms | From enrollment to the end of 12 weeks
  the changes in scores of PANSS negative subscale between the baseline and the first post-treatment measurement.

SECONDARY OUTCOMES:
congtive/negative symptoms | From enrollment to the end of 20 weeks
  the scores of MCCB/PANSS negative subscale at the eight-week follow-up after withdrawal of PQQ treatment
Malondialdehyde, Mitochondrial DNA, and Glutathione Peroxidase | From enrollment to the end of 12 weeks and 20 weeks
  The levels of biomarkers representing oxidative stress and inflammatory activity are assessed in venous blood.
Connectivity strength of target neural circuits | From enrollment to the end of 12 weeks and 20 weeks
  The functional state of target brain regions and the connectivity strength of key neural circuits, including the prefrontal-parietal cognitive control network, the hippocampal-prefrontal memory circuit, and the thalamo-cortical information gating system.

IPD SHARING:
Plan to Share IPD: Yes
required the permission from the PI
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Tamakoshi M, Suzuki T, Nishihara E, Nakamura S, Ikemoto K. Pyrroloquinoline quinone disodium salt improves brain function in both younger and older adults. Food Funct. 2023 Mar 6;14(5):2496-2501. doi: 10.1039/d2fo01515c. PMID 36807425
- [Background] Nunome K, Miyazaki S, Nakano M, Iguchi-Ariga S, Ariga H. Pyrroloquinoline quinone prevents oxidative stress-induced neuronal death probably through changes in oxidative status of DJ-1. Biol Pharm Bull. 2008 Jul;31(7):1321-6. doi: 10.1248/bpb.31.1321. PMID 18591768
- [Background] Zhang P, Xu Y, Li L, Jiang Q, Wang M, Jin L. In vitro protective effects of pyrroloquinoline quinone on methylmercury-induced neurotoxicity. Environ Toxicol Pharmacol. 2009 Jan;27(1):103-10. doi: 10.1016/j.etap.2008.08.010. Epub 2008 Sep 7. PMID 21783927
- [Background] Xiao L, Wang M, Li J, Wang H, Pu N, Bo X, Chen F, Zhou Y, Cheng Q. Pyrroloquinoline Quinone Preconditioning Alleviates Ischemic Cerebral Injury Through Antioxidant and Anti-Inflammatory Mechanisms. J Neuroimmune Pharmacol. 2025 Jul 23;20(1):75. doi: 10.1007/s11481-025-10234-1. PMID 40696055